CLINICAL TRIAL: NCT06509425
Title: Pelvic Congestion Syndrome Following Salpingectomy Compared to Tubal Ligation at Time of Caesarean Section
Brief Title: Pelvic Congestion Syndrome Post Tubal Ligation Versus Salpingectomy Performed During Caesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS 296/2024
Record Dates: First submitted 2024-04-23; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-04

CONDITIONS: Pelvic Congestion Syndrome
Keywords: salpingectomy; pelvic congestion; tubal ligation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants undergoing caesarean section and salpingectomy. (Active Comparator)
  Interventions: Procedure: salpingectomy during caesarean section
- Participants undergoing caesarean section and tubal ligation (Active Comparator)
  Interventions: Procedure: tubal ligation during caesarean section

INTERVENTIONS:
Procedure: salpingectomy during caesarean section — Salpingectomy will be done by clamping, division and ligation using adsorbable suture material (2-0 Vicryl) and excising the tube till it's isthmic part by scissors.
  Arms: Participants undergoing caesarean section and salpingectomy.
Procedure: tubal ligation during caesarean section — Tubal ligation will be done by Parkland technique. An opening is made in an avascular section of the mesosalpinx by electrocautery. Two absorbable suture ties (2-0 Vicryl) are passed through the opening and used to ligate the proximal and distal ends of the segment (at least 2 cm) which will get excised by scissors.
  Arms: Participants undergoing caesarean section and tubal ligation

SUMMARY:
Permanent tubal sterilization during Caesarean section is a reliable method of contraception. It is done either by bilateral tubal ligation or bilateral salpingectomy according to surgeon's preference.

Studies revealing bilateral salpingectomy has an added benefit of primary prevention of ovarian cancer has encouraged surgeons to perform bilateral salpingectomy rather than tubal ligation as a risk reducing surgery owing to the acceptance of fallopian tubes as the origin of high grade serous ovarian cancer.

Another aspect to take into consideration is the post tubal ligation syndrome as it severely affects the quality of life. Diagnosis is based on clinical picture, imaging, and exclusion of other causes of chronic pelvic pain. Women experience dysmenorrhea, dyspareunia, menstrual irregularities, and pelvic pain. The gold standard is venography; however, the first choice for initial evaluation is duplex ultrasound.

In this study, we assess impact of bilateral salpingectomy versus tubal ligation in terms of pelvic congestion by participant's symptoms and ultrasound findings

DETAILED DESCRIPTION:
Women planned for caesarean delivery and tubal sterilization will be screened for eligibility on presenting to the labor unit.

Informed written consent will be taken from all the participants before enrollment in the study.

Randomization will be done at a 1:1 ratio to bilateral salpingectomy or bilateral tubal ligation by a computer-generated scheme. Sequentially numbered sealed opaque envelopes will be prepared, each containing patient allocated procedure. It will be revealed to the case surgeon.

1) Surgical Intervention: Caesarean section and tubal sterilization will be performed by resident on duty.

Identification of the fimbriated end of the Fallopian tube. It will be grasped by a Babcock or Allis forceps.

Tubal ligation will be done by Parkland technique. An opening is made in an avascular section of the mesosalpinx by electrocautery. Two absorbable suture ties (2-0 Vicryl) are passed through the opening and used to ligate the proximal and distal ends of the segment (at least 2 cm) which will get excised by scissors.

Salpingectomy will be done by clamping, division and ligation using adsorbable suture material (2-0 Vicryl) and excising the tube till it's isthmic part by scissors.

Hemostasis will be ensured at the incised edges. Participants undergoing salpingectomy will have their fallopian tubes sent for pathological examination to confirm transection and exclude malignancies.

2) Postoperative assessment: Follow up visit after ten weeks.

1. History:

   The participant is asked about these symptoms:
   * Menstrual irregularities
   * Dull, noncyclical throbbing pelvic pain (unilateral or bilateral), worsened with long periods of standing or walking and punctuated by intermittent sharp pain.
2. Sonographic evaluation:

It will be done by the same investigator (Assistant Lecturer at Radiology department, Ain Shams University).

Machine used:

Samsung ultrasound machine with Transvaginal probe 5-7 Megahertz

All participants will be asked to empty their urinary bladder and will be placed in lithotomy position with adequate covering of the participants for transvaginal position. The assessment will detect:

1. Presence of pelvic varicocele. (tortuous and dilated veins that are greater than 6 mm in diameter around the ovary and uterus)
2. Maximal diameter of the pelvic venous plexus.
3. Presence of crossing veins in the myometrium.
4. Change of the duplex waveform during Valsalva's maneuver in both ovarian and internal iliac veins.

ELIGIBILITY:
Inclusion Criteria:

* Females undergoing caesarean section and requesting tubal sterilization as a permanent method of contraception.
* 30 years or older

Exclusion Criteria:

* Previous history of tubal surgery (changes in blood flow)
* Previous history of oophorectomy (changes in blood flow)
* Congenital anomalies or malformations in fallopian tubes or ovaries. (affection of normal anatomy of pelvic blood vessels)
* Women diagnosed with pelvic congestion. (Known cause for pelvic congestion other than tubal sterilization)
* High likelihood of lost to follow up.
* Inability to provide good data.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
symptoms of pelvic congestion syndrome | Ten weeks postoperative
  A questionnaire to detect changes in menstrual pattern or new onset of pelvic pain.

SECONDARY OUTCOMES:
signs of pelvic congestion syndrome | Ten weeks postoperative
  Transvaginal US will be done 10 weeks postoperative for detection of signs of pelvic congestion
intraoperative complications | intraoperative
  blood transfusion, visceral injury and increased operative time

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospitals, Cairo, Abaseya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
A case report form for each participant will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR